CLINICAL TRIAL: NCT01918644
Title: A Phase Ia-Ib Dose-escalation Study Evaluating Safety and Efficacy of Neoadjuvant Stereotactic Body Radiotherapy (SBRT) With Concomitant Capecitabine Chemotherapy for Resectable Carcinoma of Exocrine Pancreas.
Brief Title: Neoadjuvant SBRT With Concomitant Capecitabine in Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1499; NCI-2013-01347 (Registry Identifier: NCI Trial ID); 2013-0645 (Other: Institutional Review Board); RO12210 (Other: University of Wisconsin Carbone Cancer Center); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); Protocol Version 2/6/2018 (Other: UW Madison)
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Capecitabine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SBRT, capecitabine, and surgery) (Experimental): Patients undergo SBRT every other day over 2 weeks for a total of 5 fractions and receive capecitabine PO every 12 hours 5 days a week for 2 weeks. Patients then undergo definitive surgery after a minimum of 2 weeks from the completion of SBRT.
  Interventions: Radiation: stereotactic body radiation therapy; Drug: capecitabine; Procedure: therapeutic conventional surgery; Procedure: magnetic resonance imaging; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Procedure: therapeutic conventional surgery — Undergo definitive surgery
Procedure: magnetic resonance imaging — Optional correlative studies
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of stereotactic body radiation therapy when given together with capecitabine before surgery in treating patients with pancreatic cancer that can be removed by surgery. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving stereotactic body radiation therapy and capecitabine before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended-phase-II-dose (RPTD) of stereotactic body radiation therapy (SBRT) at an escalating dose schedule when combined with standard-dose capecitabine as neoadjuvant therapy for resectable carcinoma of exocrine pancreas.

SECONDARY OBJECTIVES:

I. To estimate the incidence of overall 30-day post-operative complications.

II. To estimate the radiological response rates.

III. To estimate the pathological response rates.

IV. To estimate the rates of resection with negative margins.

V. To estimate the recurrence free survival (RFS).

VI. To estimate the overall survival (OS).

TERTIARY OBJECTIVES (OPTIONAL):

I. To define tumor volume (TV), dynamic contrast enhancement (DCE) pattern and mean apparent diffusion coefficient (ADC) measurements in diffusion-weighted magnetic resonance (MR) imaging (DWI) in patients with resectable pancreatic cancer undergoing neoadjuvant SBRT and concomitant chemotherapy (ChT).

II. To correlate TV, DCE and ADC measurements at baseline magnetic resonance imaging (MRI) versus final pathological response.

III. To correlate TV, DCE and ADC changes from baseline in MRI done three weeks post-SBRT versus final pathological response.

IV. To predict surgical margin status using MRI done at baseline and at three weeks post-SBRT.

V. To correlate TV, DCE and ADC changes from baseline in MRI done post-3rd fraction at baseline versus final pathological response.

VI. To describe in the biopsy and/ or the surgical specimen, expression of following markers: secreted protein acidic and rich in cysteine (SPARC) expression; distribution of pancreatic stellate cells (PSC); distribution of cluster of differentiation (CD)4+/ CD8+ T cell, CD56+ natural killer (NK) cells; other molecular and inflammatory cellular markers may be explored.

VII. To describe changes induced by neoadjuvant therapy by comparison of expression of these markers between the biopsy and the surgical specimen.

VIII. To compare baseline and/ or post-treatment expression with treatment response, toxicity and clinical survival outcome.

OUTLINE: This is a dose-escalation study of SBRT.

Participants undergo SBRT every other day over 2 weeks for a total of 5 fractions and receive capecitabine orally (PO) every 12 hours 5 days a week for 2 weeks. Participants then undergo definitive surgery after a minimum of 2 weeks from the completion of SBRT.

After completion of study treatment, participants are followed up at 1 month and 3 months, every 3 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of exocrine pancreatic head amenable to oncological surgical resection per findings on a pancreatic-specific computed tomography (CT) or MRI scan. Tumors of the body that allow a surgical approach similar to pancreatic head tumors are acceptable.
* Must be deemed a surgical candidate by the surgical oncology service.
* Eastern Cooperative Oncology Group (ECOG) performance score of =< 2
* Signed informed consent document(s)
* Patients with no evidence of regional or distant metastatic disease based on CT scan of the chest/ abdomen/pelvis.
* Absolute neutrophil count (ANC) >= 1,500 cells/mm3
* Platelet count >= 100,000 cells/mm3
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 times the upper limit of normal
* Total bilirubin =< 3 times the upper limit of normal if patient had recent biliary stenting, total bilirubin =< 1.5 times the upper limit of normal if no biliary stenting was done
* Serum creatinine within normal range with a creatinine clearance >= 30 ml/min
* Neoadjuvant chemotherapy will be permitted prior to the initiation of SBRT radiation therapy on this clinical trial. There must be a minimum of 2 weeks between the completion of any neoadjuvant chemotherapy and the beginning of SBRT radiation therapy. Furthermore, restaging must be done prior to registration to ensure that patients remain resectable.

Exclusion Criteria:

* Patients with primary ampullary, biliary or duodenal cancer would be excluded
* Patients with tumors primarily of the body or tail of the pancreas requiring a distal pancreaticoduodenectomy would be excluded
* (H/ o) Crohn's disease/ ulcerative colitis/ scleroderma
* History of prior allergic reactions attributed to compounds of similar chemical or biologic composition as capecitabine
* History of prior allergic reactions attributed to compounds of CT/ MRI contrast that cannot be managed with appropriate pre-medication prophylaxis and thereby preclude use of baseline/ follow-up or radiation planning imaging
* Any prior external beam radiation will be evaluated to determine radiation field overlaps and appropriateness of protocol radiation, any invasive cancer in the last 5 years (except for a diagnosis of low-risk prostate cancer, treated non-melanoma/melanoma skin cancer, appropriately treated ductal carcinoma in situ or early stage invasive carcinoma of breast and appropriately treated in-situ/early stage cervical/endometrial cancer)
* Pregnant or nursing women; women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the point of study entry and for the duration of all active treatments; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Treatment with a non-approved or investigational drug within 28 days of study treatment
* History of having MRI non-compatible metal (injury- or treatment-related) in the body will be an exclusion criteria specific to the MRI sub-study
* Considering the small size of the PET/MR scanner bore, subjects with known severe claustrophobia or with body habitus not compatible with the bore (>300lbs, BMI>40) may also have to be excluded.
* Subjects unable to maintain blood glucose less than 200mg/dl may not be suitable for the PET/MRI substudy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity defined as any grade 3-4 non-hematologic toxicity or grade 5 toxicity attributable to combination chemo-radiotherapy per the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 90 days from the start of SBRT and capecitabine
  The number and percent of patients reporting adverse events (all, severe or worse, serious and related) will be quantified for each dose level.

SECONDARY OUTCOMES:
Incidence of 30-day post-operative complications | 30 days
  Will be expressed as a percentage.
Radiological response per Response Evaluation Criteria in Solid Tumors (RECIST) and volumetric measurements | Up to 3 years
  Will be expressed as a percentage.
Pathological response, graded based on the College of American Pathologists (CAP) and Ishikawa, Evans, and Chun grading systems | Up to 3 years
  Will be expressed as a percentage.
Incidence of margin-negative resection, defined as the absence of viable tumor cells at the inked surgical margin | Up to 3 years
  Will be expressed as a percentage.
Loco-regional recurrence free survival, defined with follow-up radiological assessment | From the point of start of SBRT to the point of recurrence or death, assessed up to 3 years
  Kaplan-Meier estimates will be calculated. Log-rank test and Cox regression analysis will be used for univariate and multivariate analyses, respectively. Chi square and regression analysis will be performed to test association of categorical variables with treatment response.
OS | From the point of start of SBRT to the time of death or last follow-up if alive, assessed up to 3 years
  Kaplan-Meier estimates will be calculated. Log-rank test and Cox regression analysis will be used for univariate and multivariate analyses, respectively. Chi square and regression analysis will be performed to test association of categorical variables with treatment response.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bassetti, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/